CLINICAL TRIAL: NCT04520100
Title: Pilot Trial of Hypnosis and Enhanced Communication Training to Reduce Anxiety, Improve Patient Satisfaction, and Decrease Movement for Patients Undergoing Magnetic Resonance Imaging
Brief Title: Pilot Trial of Hypnosis and Enhanced Communication In Patients Undergoing MRI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Prevention
Other Study IDs: 20-1576
Record Dates: First submitted 2020-07-31; First posted 2020-08-20 (Actual); Last update posted 2022-05-05 (Actual); Status verified 2022-05

CONDITIONS: Claustrophobia; Anxiety; Magnetic Resonance Imaging
MeSH Terms: conditions — Claustrophobia; Anxiety Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- MRI without intervention (No Intervention): No hypnosis during MRI and care by regular MR technologist
- MRI with clinical hypnosis and regular MR tech (Active Comparator): Hypnosis during MRI and care by regular MR technologist
  Interventions: Behavioral: Clinical Hypnosis performed by the PI
- MRI with care by MR Tech trained in empathic communication (Active Comparator): No hypnosis during MRI and care by MR technologist who have been trained in emphatic communication
  Interventions: Behavioral: Care by technician trained in empathic communication

INTERVENTIONS:
Behavioral: Clinical Hypnosis performed by the PI — The patient will receive clinical hypnosis by the PI prior to examination and listen to recorded session during their MRI.
  Arms: MRI with clinical hypnosis and regular MR tech
Behavioral: Care by technician trained in empathic communication — The patient will be taken care of by an MRI technician who has been previously trained in empathic communication.
  Arms: MRI with care by MR Tech trained in empathic communication

SUMMARY:
The overarching goal of this study is to enhance patient comfort during magnetic resonance (MR) exams by reducing anxiety and movement during the exam, thereby decreasing the time spent in magnetic resonance imaging (MRI) scanner and potentially improving patient satisfaction with the clinical care experience. This will be done with a trial focusing on studying the effects of clinical hypnosis and focused communication training on patient anxiety and other metrics during an MRI examination.

DETAILED DESCRIPTION:
Magnetic resonance imaging (MRI) is an increasingly common imaging modality used for the diagnosis and treatment of disease. Given the closed bore nature of the MRI machine itself, the need to hold still within the imaging bore, the high noise level, vibrations and other uncomfortable sensations that can be experienced during MRI, anxiety and other claustrophobia-related symptoms are relatively frequently reported . These symptoms may result in premature termination/failure of the MRI examination, or excessive patient movement which can degrade image quality and lengthen the time needed to perform the examination. Additionally, patient satisfaction scores suffer due to these negative experiences during MRI. This is especially important, as radiology departments are major influencers in overall hospital patient satisfaction scores .

Due to the substantial impact that anxiety and claustrophobia-related symptoms have on all aspects of MRI, the most common intervention provided to patients who report such symptoms are anxiolytic medications or sedation/anesthesia. These interventions can come at significant cost to patients and radiology departments and carry medical risks to the patient as well. Anxiolytic medications or sedation/anesthesia can lead to potential negative side effects, such as cardiopulmonary depression, hypotension, tachycardia, dystonic reactions, involuntary muscle movements . These adverse effects can even contribute to unsuccessful imaging themselves.

Non-medical interventions, such as clinical hypnosis and enhanced communication strategies are not well studied in MR and have the potential to provide similar benefits of anxiolytic medications or sedation in terms of reducing movement artifacts and anxiety, but with far fewer side effects and safety concerns. For example, hypnosis can reduce anxiety and operating room time during radiological procedures , reduce amounts of analgesic used , and decrease behavioral issues related to claustrophobia during MRI . Additionally, enhanced communication strategies can reduce MRI no-show and study failure rates and improve ratings in national Hospital Consumer Assessment of Healthcare Providers and Systems (HCAHPS) .

Thus, there is evidence to support the use of hypnosis and communication training during MRI in order to improve MR exam outcomes and patient outcomes.

The investigators hypothesis is that patients who participate in hypnosis prior to MRI will experience less anxiety and demonstrate less movement during the exam. This will lead to improved overall patient satisfaction, reduction in image repeat rates and the overall time needed to perform the MRI.

The investigators also hypothesize that patients who undergo MRI with a radiology technician who has received training in enhanced communication skills will experience less anxiety and demonstrate less movement during the exam. This will lead to improved overall patient satisfaction and reduction in image repeat rates and the overall time needed to perform the MRI.

ELIGIBILITY:
Inclusion Criteria:

* Patients over 18 years old, undergoing MRI at the UCH Outpatient Pavilion.
* Are scheduled to undergo an MRI that does not require deep breath holds
* English-speaker

Exclusion Criteria:

* Patients under the age of 18 years old,
* Diagnosis of active psychosis,
* Diagnosis of delirium
* Diagnosis of movement disorders
* Those who lack mental capacity to complete the forms.
* Scheduled to undergo MRI with deep breath holds.
* Non-English speaker

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2020-10-02 (Actual); Primary Completion 2022-01-23 (Actual); Study Completion 2022-01-23 (Actual)

PRIMARY OUTCOMES:
State and Trait Anxiety Inventory for Adults (STAI-AD) (Pre-MRI) | Just prior to MRI on the same day as the MRI examination
  Patient will complete the STAI-AD Short forms. Higher scores are correlated with higher anxiety (a worse outcome) and lower scores are correlated with less anxiety. Maximum score is 80 and minimum score is 20.
State and Trait Anxiety Inventory for Adults (STAI-AD) (Post-MRI) | Immediately after MRI
  Patient will complete the STAI-AD Short forms. Higher scores are correlated with higher anxiety (a worse outcome) and lower scores are correlated with less anxiety. Maximum score is 80 and minimum score is 20.
Patient Satisfaction Inventory | Immediately after MRI
  Patient will complete the patient satisfaction survey.

SECONDARY OUTCOMES:
Movement/Image Repeat Rate | During the MRI examination
  MRI technician will record the number of repeated acquisitions needed during the MRI exam.
Length of MRI examination | During the MRI examination
  Length of MRI from 1st image to last image obtained will be obtained from the medical record.
Pulse Oximetry Vales | During the MRI examination.
  Patient's pulse oximetry values will be measured throughout the MRI .

CONTACTS AND LOCATIONS:
Overall Officials: Alexandra Chadderdon, PsyD, Principal Investigator — University of Colorado Denver, Anschutz Medical Campus
Locations (1):
- University of Colorado Anschutz Medical Campus, Aurora, Colorado, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lang EV, Yuh WT, Ajam A, Kelly R, Macadam L, Potts R, Mayr NA. Understanding patient satisfaction ratings for radiology services. AJR Am J Roentgenol. 2013 Dec;201(6):1190-5; quiz 1196. doi: 10.2214/AJR.13.11281. PMID 24261356
- [Background] Norbash A, Yucel K, Yuh W, Doros G, Ajam A, Lang E, Pauker S, Mayr N. Effect of team training on improving MRI study completion rates and no-show rates. J Magn Reson Imaging. 2016 Oct;44(4):1040-7. doi: 10.1002/jmri.25219. Epub 2016 Apr 6. PMID 27126735
- [Background] Simon EP. Hypnosis using a communication device to increase magnetic resonance imaging tolerance with a claustrophobic patient. Mil Med. 1999 Jan;164(1):71-2. PMID 9922650

DOCUMENTS (1):
  • Informed Consent Form (2020-07-14): https://cdn.clinicaltrials.gov/large-docs/00/NCT04520100/ICF_000.pdf